CLINICAL TRIAL: NCT02438761
Title: Phase II Evaluating the Efficacy of the Dual Inhibition of Phosphoinositide 3 Kinase (PI3K)/Akt /Mammalian Target Of Rapamycine (mTOR) Signaling Pathway by PF-05212384 (PKI-587) for Patients With Myeloid Neoplasm Secondary to Chemo-radiotherapy (t-AML/MDS) or de Novo Relapsed or Refractory AML.
Brief Title: PF-05212384 (PKI-587) for t-AML/MDS or de Novo Relapsed or Refractory Acute Myeloid Leukemia (AML) (LAM-PIK)
Acronym: 5
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No objective response was observed at the first step. The treatment was considered ineffective, with a complete clinical trial suspension.
Sponsor: Institut Curie (Other)
Collaborators: Fondation ARC (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2014-10
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2019-02

CONDITIONS: Therapy-related Acute Myeloid Leukemia and Myelodysplastic Syndrome; Acute Myeloid Leukemia, in Relapse; de Novo Acute Myeloid Leukemia at Diagnostic
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndrome; PIK/Akt/mTor
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — gedatolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-05212384 (Experimental): 150 mg Intra-venous every week
  Interventions: Drug: PF-05212384

INTERVENTIONS:
Drug: PF-05212384 — PF-05212384 will be delivered by intra-venous route at a fixed dose of 150 mg per week. Each treatment cycle includes four weekly injections
  The treatment is administered in cycles of 28 days for a period of 4 cycles. Patients will be treated on a weekly basis continuously during 112 days or until progression.
  Other Names: PKI-587

SUMMARY:
Phase II open-label single-arm prospective multicentric clinical trial of PF-05212384 (PKI-587) delivered by intravenous route. A 2-stage Fleming design will be employed.

DETAILED DESCRIPTION:
The treatment is administered in cycles of 28 days for a period of 4 cycles. Patients will be treated on a weekly basis continuously during 112 days or until progression.

Blood tests (hemogram) are assessed weekly before each injection of PF-05212384 (PKI-587). Bone marrow aspiration (myelogram) is performed to evaluate the response before starting treatment and before the start of cycle 3 (after two cycles) and at the end of the study (after four cycles). Good responders who continue treatment after four cycles will be evaluated by bone marrow aspiration (myelogram) every two cycles and after the end of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patients belong to one of three categories:

   * Myeloid neoplasm secondary to chemo-radiotherapy (t-AML/MDS) aged 60 and over with unfavorable cytogenetics (European Leukemia Network definition 2010), the first cancer must have been in remission for more than two years, except in situ carcinoma, basal cell carcinoma and squamous cell carcinoma
   * Relapsed or refractory de novo AML aged 18 and over (multiple relapses allowed), regardless of the risk group, provided not being eligible for allogeneic bone marrow transplantation
   * de novo AML at diagnosis, aged 60 and over and considered unfit to benefit from induction chemotherapy associated with aplasia (at the discretion of the investigator)
2. Adequate glycemic balance defined by glycated hemoglobin ≤ 8%
3. Females of childbearing potential (FCBP) should receive effective contraception: a negative pregnancy blood test is required within 2 weeks before starting experimental treatment.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2
5. Absence of severe or active infection
6. Adequate systolic cardiac function : Left Ventricular Ejection Fraction (LVEF) ≥ 50%
7. Adequate hepatic function: Aspartate Aminotransferase Test (AST) and Alanine Aminotransferase Test (ALT) ≤ 3 times the upper limit of normal (ULN), bilirubin ≤ 1.5 x ULN
8. Adequate renal function: serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance > 60 ml/min.
9. Signed informed consent

Exclusion Criteria:

1. Glucose intolerance or diabetes mellitus, treated or untreated
2. First cancer in evolution(solid tumor or lymphoma) or in remission for less than two years, except in situ carcinoma, basal cell carcinoma and squamous cell carcinoma
3. AML secondary to MDS or myeloproliferative syndrome (WHO 2008 definitions)
4. Acute Promyelocytic Leukaemia (APL or AML French American British (FAB) classification 3) de novo or secondary to treatment (t-APL)
5. de novo or secondary Core Binding Factor (CBF)/AML
6. de novo or secondary Philadelphia Chromosome (Ph) 1 positive AML defined by the presence of a t(9.22) or a Breakpoint Cluster Region-Abelson Murine Leukemia Viral Oncogene Homolog (BCR-ABL) transcript
7. Leukocytes above 30.000/mm3 (30 G/L) at enrollment
8. Antileukemic treatment within 15 days before enrollment, with the exception of hydroxyurea
9. Central nervous system leukemic involvement
10. Pregnant or lactating women, or women of childbearing potential without effective contraception
11. Prior history of allogeneic bone marrow transplantation
12. Prior history of organ transplantation or other cause of severe or chronic immunodeficiency Human
13. Seropositivity for Human Immunodeficiency Virus (HIV) or Human T-Lymphotropic Virus-1 (HTLV-1) viruses, active B or C hepatitis
14. Inclusion in another experimental anti-cancer clinical trial*
15. Patients unable to undergo medical monitoring for geographical, social or psychological issues
16. Patient under measure of legal protection
17. No social security

    * For ethical reasons, the exclusion period before considering the possibility of participating in another clinical study with a new experimental molecule cannot be determined, yet each case will be discussed on an individual basis with the study coordinator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of PF-05212384 | 4 months after treatment
  The overall response rate will be assessed according to the International Working Group (IWG) AML and MDS criteria (by B.D. Cheson).

SECONDARY OUTCOMES:
Tolerance and toxicity during treatment | 4 months
  Issued the Common Terminology Criteria for Adverse Events (CTCAE) version 4 National Cancer Institute (NCI)
Treatment compliance | 4 months
  Treatment compliance will be assessed by the ratio between the number of cycles administered on the expected number of cycles, and on time between treatment cycles
Progressive Free Survival (PFS) | one year
  Progressive Free Survival at one year from the date of inclusion to the date of progression of the disease or death
Overall survival | 48 months
  Overall Survival from the date of inclusion to the date of death
Evaluation of Quality of life | 4 months
  Quality of life (QLQ-C30) questionnaire according to European Organisation for Research and Treatment of Cancer (EORTC)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Vargaftig, MD, Principal Investigator — Institut Curie - Hôpital René Huguenin
Locations (5):
- France (5):
  - CHU de Toulouse, Toulouse, Midi-Pyrénées
  - Institut Paoli Calmette, Marseille, PACA
  - Hôpital Saint-Louis, Paris, Île-de-France Region
  - Hôpital Cochin, Paris, Île-de-France Region
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud, Île-de-France Region